CLINICAL TRIAL: NCT02244606
Title: Open-Label, Randomized Study to Estimate Safety, PK, and Efficacy of Oral Ibrexafungerp (SCY-078) vs. Standard-of-Care Following IV Echinocandin Therapy in the Treatment of Invasive Candidiasis in Hospitalized Nonneutropenic Adults
Brief Title: Oral Ibrexafungerp (SCY-078) vs Standard-of-Care Following IV Echinocandin in the Treatment of Invasive Candidiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCY-078-202
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Mycoses; Candidiasis, Invasive; Candidemia
Keywords: Invasive Candidiasis; Invasive Candida infections; Candidemia; SCY-078; Micafungin; Fluconazole; Echinocandin
MeSH Terms: conditions — Mycoses; Candidiasis, Invasive; Candidemia | interventions — ibrexafungerp; Fluconazole; Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SCY-078 500 mg (Experimental): A single loading dose of SCY-078 1000-mg orally on the first day, followed by SCY-078 500-mg orally once-daily on subsequent days.
  Interventions: Drug: SCY-078
- SCY-078 750 mg (Experimental): A single loading dose of SCY-078 1250-mg orally on the first day, followed by SCY-078 750-mg orally once-daily on subsequent days.
  Interventions: Drug: SCY-078
- Standard-of-care (Active Comparator): Oral fluconazole 400 mg daily (with a loading dose of 800 mg on the first day) or IV micafungin 100 mg daily.
  Interventions: Drug: Fluconazole; Drug: Micafungin

INTERVENTIONS:
Drug: SCY-078
  Arms: SCY-078 500 mg; SCY-078 750 mg
Drug: Fluconazole
  Arms: Standard-of-care
Drug: Micafungin
  Arms: Standard-of-care

SUMMARY:
The purpose of this study is to compare the safety, pharmacokinetics, and efficacy of oral SCY-078 vs. standard-of-care following initial intravenous echinocandin therapy in the treatment of invasive candidiasis.

DETAILED DESCRIPTION:
Patients will receive initial intravenous (IV) echinocandin therapy. Patients who are eligible for randomization will receive SCY-078 500-mg orally, SCY-078 750-mg orally, or standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive candidiasis defined as a positive culture of blood or from another normally sterile site for Candida.
* Not of reproductive potential or if of reproductive potential, agrees to remain abstinent or use 2 methods of contraception.

Exclusion Criteria:

* Patient with Candida endocarditis, osteomyelitis, meningitis, or chronic disseminated candidiasis or evidence of endophthalmitis.
* Patient has failed treatment with an echinocandin for this episode of invasive candidiasis.
* Infection limited to the oropharynx, esophagus, urogenital system, or skin, or sputum/bronchoalveolar lavage culture.
* Participation in a clinical study with other investigational drug(s) within 30 days prior to study entry or during this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (30):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Georgia Regents University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Albany Medical Center, Albany, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - South Texas Veterans Healthcare System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
- El Salvador (2):
  - Hospital Militar Central, San Salvador
  - Hospital Rosales, San Salvador
- University of Cologne, Cologne, North Rhine-Westphalia, Germany
- Finca El Palomar, Guatemala City, Guatemala
- Honduras (2):
  - Hospital Mario Catarino Rivas, San Pedro Sula, Cortés Department
  - Instituto Hondureno de Seguridad Social Sucursal San Pedro Sula, San Pedro Sula, Cortés Department

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled, two of whom failed to meet all inclusion and exclusion criteria and were considered screen failures. Among the 25 enrolled participants who met all inclusion and exclusion criteria, three were not randomized. Thus, 22 patients were randomized to receive SCY-078 500 mg or SCY-078 750 mg or standard-of-care.
Groups:
- Ibrexafungerp 500-mg: A single loading dose of SCY-078 1000-mg orally on the first day, followed by SCY-078 500-mg orally once-daily on subsequent days.
- Ibrexafungerp 750-mg: A single loading dose of SCY-078 1250-mg orally on the first day, followed by SCY-078 750-mg orally once-daily on subsequent days.
- Standard of Care (Fluconazole): Oral fluconazole 400 mg daily (with a loading dose of 800 mg on the first day
- Standard of Care (Micafungin): IV micafungin 100 mg daily
Period: Overall Study
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Started | 7 | 7 | 7 | 1
Did Not Receive Study Drug | 1 | 0 | 0 | 0
Did Not Complete Randomized Study Drug | 1 | 1 | 2 | 0
Completed | 4 | 2 | 4 | 0
Not Completed | 3 | 5 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Did Not Complete Study for Reason Other: | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 1 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 1 | 19
  >=65 years | 1 | 1 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (7.81) | 48.9 (15.46) | 49.6 (15.66) | 63.0 (NA) — SD was not estimated because only one participant was analyzed. | 52.1 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 0 | 11
  Male | 5 | 3 | 2 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 7 | 6 | 1 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 4 | 6 | 6 | 1 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability, Assessed by Adverse Events, Clinical Laboratory Results, Physical Examination Findings, ECG Results, and Vital Sign Measurements
Description: All Related TEAEs by SOC and PT, by Treatment, Safety
Time Frame: up to 10 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Number analyzed (Participants) | 6 | 7 | 7 | 1
Participants
  Patients with at least One Drug-Related TEAE | 1 | 1 | 0 | 0
  Patients with no Drug- Related TEAE | 5 | 6 | 7 | 1

2. Primary Outcome: Dose of SCY-078 That Achieves the Target Exposure (AUC)
Description: Summary of PK Parameters on Day 1 by Treatment Arm, from non-compartmental analysis, PK
Time Frame: 0 to 24 hours post-dose
Population: Pharmacokinetic Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg
Number analyzed (Participants) | 5 | 5
Participants | 3 | 4

3. Secondary Outcome: Global Response
Description: Participant's clinical response (signs or symptoms) and microbiological response (presence of Candida culture)
Time Frame: end of all antifungal therapy (administered for a maximum of 28 days)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Number analyzed (Participants) | 7 | 7 | 7 | 1
Participants
  Favorable | 5 | 6 | 5 | 1
  Unfavorable | 2 | 1 | 2 | 0

4. Secondary Outcome: Clinical Response
Description: Participant's persistence of signs or symptoms and administration of systemic non-study antifungal therapy
Time Frame: end of all antifungal therapy (administered for a maximum of 28 days)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Number analyzed (Participants) | 7 | 7 | 7 | 1
Participants
  Favorable | 5 | 6 | 5 | 1
  Unfavorable | 1 | 0 | 2 | 0
  Unknown | 1 | 1 | 0 | 0

5. Secondary Outcome: Microbiological Response
Description: Cultures or radiographs/imaging of blood or non-blood sites of infection showing evidence of Candida infection
Time Frame: end of all antifungal therapy (administered for a maximum of 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Number analyzed (Participants) | 7 | 7 | 7 | 1
Participants
  Favorable | 6 | 6 | 6 | 1
  Unfavorable | 0 | 0 | 1 | 0
  Unknown | 1 | 1 | 0 | 0

6. Secondary Outcome: Relapse
Description: If Invasive Candida infection recurs or if antifungal therapy for a proven or suspected Candida infection is administered
Time Frame: 2 weeks and 6 weeks after the end of all antifungal therapy, up to 10 weeks
Population: Intent-To-Treat (ITT): All randomized participants
  Overall number of participants includes all randomized participants, number analyzed includes participants analyzed at a particular time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
Number analyzed (Participants) | 7 | 7 | 7 | 1
Participants
  Week 2 Post-Treatment: Relapsed | 1 | 0 | 0 | 0
  Week 2 Post-Treatment: Did Not Relapse | 4 | 4 | 5 | 0
  Week 2 Post-Treatment: Not Evaluable or Missing | 2 | 3 | 2 | 1
  Week 6 Post-Treatment: Relapsed | 0 | 0 | 0 | 0
  Week 6 Post-Treatment: Did Not Relapse | 4 | 2 | 4 | 0
  Week 6 Post-Treatment: Not Evaluable or Missing | 3 | 5 | 3 | 1

ADVERSE EVENTS:
Arm/Group | Ibrexafungerp 500-mg | Ibrexafungerp 750-mg | Standard of Care (Fluconazole) | Standard of Care (Micafungin)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/7 | 1/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/7 | 3/7 | 0/1
Other Adverse Events (participants affected / at risk) | 5/6 | 4/7 | 4/7 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp 500-mg (N=6) | Ibrexafungerp 750-mg (N=7) | Standard of Care (Fluconazole) (N=7) | Standard of Care (Micafungin) (N=1)
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 0
Bacteremia (Infections and infestations) | 1 | 0 | 0 | 0
Fungemia (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute lymphocytic leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp 500-mg (N=6) | Ibrexafungerp 750-mg (N=7) | Standard of Care (Fluconazole) (N=7) | Standard of Care (Micafungin) (N=1)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No